CLINICAL TRIAL: NCT05558241
Title: Micro-UltraSound In Cancer - Active Surveillance (MUSIC-AS)
Brief Title: Micro-UltraSound In Cancer - Active Surveillance
Acronym: MUSIC-AS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HREBA.CC-22-0135
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: Active surveillance; micro-ultrasound
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective paired diagnostic trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combined MRI and micro-ultrasound guided prostate biopsy. (Experimental): In a single biopsy session, first, a microUS-guided biopsy of regions of interest (ROIs) will be performed. The MRI fusion software will then be turned on, the clinician unblinded to the MRI results, and biopsy cores from within the boundaries of the MRI-fused lesion will be sampled from ROIs. Up to two ROIs identified on microUS or MRI will be targeted with up to 3 cores per ROI. If the MRI ROIs overlap with the microUS ROIs after unblinding, then the cores taken during the microUS-guided biopsy will be counted as both microUS and MRI-guided. Finally, a standard 12-core systematic biopsy will be performed.
  Interventions: Device: High-resolution micro-ultrasound

INTERVENTIONS:
Device: High-resolution micro-ultrasound — In a single biopsy session, first, a microUS-guided biopsy of regions of interest (ROIs) will be performed. The MRI fusion software will then be turned on, the clinician unblinded to the MRI results, and biopsy cores from within the boundaries of the MRI-fused lesion will be sampled from ROIs. Up to two ROIs identified on microUS or MRI will be targeted with up to 3 cores per ROI. If the MRI ROIs overlap with the microUS ROIs after unblinding, then the cores taken during the microUS-guided biopsy will be counted as both microUS and MRI-guided. Finally, a standard 12-core systematic biopsy will be performed.

SUMMARY:
This study will compare the two imaging modalities (MRI and micro-ultrasound) during Active Surveillance of prostate cancer (PCa). Progression to clinically significant PCa will be assessed by first taking micro-US targeted samples (while blinded to MRI results), followed by MRI targeted samples, finishing with 12 systematic biopsy cores. The primary goal is to compare microUS to MRI for the detection of ≥GG2 PCa at confirmatory biopsy. This study will also collect blood samples from participants to be used for future biomarker studies.

ELIGIBILITY:
Inclusion Criteria:

* Adult men with Gleason Grade Group 1 prostate cancer managed by active surveillance who require a confirmatory prostate biopsy

Exclusion Criteria:

* Men who cannot undergo a prostate MRI
* Men who cannot undergo a prostate biopsy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 210 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2033-06-30 (Estimated)

PRIMARY OUTCOMES:
Cancer upgrading during Active surveillance by micro-ultrasound and MRI | Immediately after biopsy.
  The primary outcome will be detection of ≥Grade Group 2 by each biopsy, technique in combination with the systematic biopsy.

SECONDARY OUTCOMES:
Cancer upgrading during Active surveillance between imagine-guided versus systematic biopsy. | Immediately after biopsy.
  Secondary outcome will compare each imaged-guided biopsy technique to the standard-of-care 12 core systematic biopsy simultaneously obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Kinnaird, MD, PhD, Principal Investigator — University of Alberta
Locations (5):
- University of California Los Angeles, Department of Urology, Los Angeles, California, United States
- Canada (3):
  - Kipnes Urology Centre - Kaye Edmonton Clinic, Edmonton, Alberta
  - University of British Columbia, Vancouver, Alberta
  - CIUSSS du Nord-de-L'Ile-De-Montreal, Montreal, Quebec
- Humanitas, Milan, Italy